CLINICAL TRIAL: NCT05740943
Title: Induction Lorlatinib for ALK Fusion Locally Advanced Non-small Cell Lung Cancer: A Prospective, Single Arm, Open-label Phase 2 Study
Brief Title: Induction Lorlatinib in Stage III Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: Guangzhou No.12 People's Hospital (Other Government); Peking Union Medical College Hospital (Other); Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Wen-zhao ZHONG, Head of Pulmonary Surgery, Guangdong Provincial People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LORIN
Record Dates: First submitted 2023-02-12; First posted 2023-02-23 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Stage III NSCLC; Surgery
Keywords: ALK fusion; Induction Treatment; Multidisciplinary; ctDNA; Lorlatinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — lorlatinib

STUDY DESIGN:
Intervention Model Description: A Simon two-stage design was applied. Primary endpoint for this study was pCR. The unacceptable response rate for pCR was less than 20% and desirable response rate was 40%. The error rate for alpha was set as 0.05 and 0.2 for beta. The Optimal assay was chosen and 43 patients were to be enrolled to meet adequate statical power. 13 patients would be enrolled in stage I and at least 3 patients achieved pCR were required to proceed stage II enrollment. Overall, if 12 patients achieved pCR, the study would be determined as positive. 10% drop-off rate should be considered and at least 48 patients should be enrolled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Patients will receive 12-week induction Lorlatinib followed by radical surgery or local radiotherapy or continue Lorlatinib through MDT and optional consolidation lorlatinib for up to 2 years.
  Interventions: Drug: Lorlatinib

INTERVENTIONS:
Drug: Lorlatinib — Patients were assigned to receive oral lorlatinib at a dose of 100 mg daily in a course of treatment that was measured in cycles of 28 days. 3 cycles of induction treatment will be required for the study.

SUMMARY:
A prospective, single-arm, open-label phase 2 study that evaluates the efficacy and safety of induction Lorlatinib in stage III non-small cell lung cancer and explores the clinical feasibility of dynamic ctDNA and multidisciplinary assessment in guiding local treatments.

DETAILED DESCRIPTION:
Simon two-stage was applied to estimate the required sample size for the study. Overall an estimated 43 patients were required and at least 12 patients achieved pathological complete response would be deemed as positive result. Patients will be provided 3 cycles induction Lorlatinib 100mg and then assessed whether patients would be eligible for radical surgery or local radiotherapy through multidisciplinary evaluation. After local intervention, patients could choose consolidation treatment of Lorlatinib for up to 2 years or adjuvant doublet chemotherapy for up to 4 cycles. Dynamic blood samples will be collected before and after induction Lorlatinib as well as consolidation treatment. The primary endpoints is pCR for patients who received radical surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age :18 Years to 75 Years;
* ECOG physical score 0-2 points; expected survival time ≥ 1 year;
* Pathologically confirmed diagnosis with Stage III NSCLC which harbored ALK fusion detected by next generation sequencing (NGS) or immunohistochemistry (IHC) with or without FISH. Suspected N2 (station 2/4/7) for stage III disease should be confirmed by either mediastinoscopy or EBUS.
* At least one measurable target lesion according to the RECIST 1.1 standard;
* The main organ function meets the following criteria: 1) blood routine: absolute value of neutrophils ≥ 1.5 × 109 / L, platelets ≥ 75 × 109 / L, hemoglobin ≥ 80 g / L; 2) blood biochemistry: total bilirubin ≤ 1.5 times the upper limit of normal value, aspartate aminotransferase and alanine aminotransferase ≤ 2.5 times the upper limit of normal value (if liver metastasis, ≤ upper limit of normal value 5 times), serum creatinine ≤ 1.5 times the upper limit of normal;
* Subjects voluntarily joined the study and signed informed consent, with good compliance to follow-up.

Exclusion Criteria:

* Stage I, stage II and metastatic stage IV NSCLC;
* Histologically confirmed small cell lung cancer (including lung cancer mixed with small cell lung cancer and non-small cell lung cancer);
* Patients who have previously used any other anti-tumor drugs or received surgery/radiotherapy;
* Patients with any underlying disease that investigators consider it may affect patient's prognosis including sever cardiovascular, pulmonary disease or serious infections.
* Clinically obvious gastrointestinal abnormalities, which may affect the intake, transport or absorption of drugs (such as inability to swallow, chronic diarrhea, intestinal obstruction, etc.), or patients with total gastrectomy;
* Pregnant or lactating women; those who have fertility are unwilling or unable to take effective contraceptive measures;
* Patients with low compliance or willingness to take the drugs and surveillance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) | After surgery (approximately 2 weeks)
  The pathological complete response is defined as the absence of residual tumor in both lung and regional lymph nodes after induction treatment and radical surgery.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | From date of induction treatment till the date of first documented disease progression or death, whichever came first, assessed up to 48 months
  The period after initiation of induction treatment till the time of disease progress or any cause of death.
Objective Response Rate (ORR) | After last dose of induction treatment (approximately 1 week)
  ORR is the number of participants with a Complete Response (CR) and Partial Response (PR) divided by the total number of enrolled participants per arm, then multiplied by 100. Response is based on the Response Evaluation Criteria In Solid Tumors (RECIST 1.1) criteria. Complete Response (CR) was defined as the disappearance of all target lesions. Partial Response (PR) was defined as at least a 30% decrease in sum of longest diameter of target lesions compared to baseline or the complete disappearance of target lesions, with persistence of 1 or more nontarget lesion(s) and no new lesions.
Event-free Survival (EFS) | From date of radical surgery till the date of first documented disease relapse, assessed up to 48 months
  The period after radical surgery till the time of disease relapse with either local recurrence or distant metastasis.
Dynamic ctDNA alteration | From induction treatment till completion of consolidation lorlatinib (approximately 2.5 years)
  The exploratory ctDNA alteration will be stratified into three parts. 1) Induction period: overall ctDNA clearance rate (before and after induction treatment); 2) Posttreatment period: ctDNA clearance rate after local treatment; 3) Consolidation period: 1-year and 2-year ctDNA positive rate during consolidation treatment.
Overall Survival (OS) | From date of induction treatment till the date of death from any cause, assessed up to 60 months.
  OS was assessed from initiation of treatment to death as a result of any cause.
Adverse Events (AEs) | From Initiation of induction treatment till treatment discontinuation, assessed up to 24 months.
  Incidence of AE/SAE which has been confirmed correlation with Lorlatinib or local treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Zhao Zhong, MD., Principal Investigator — Guangdong Provincial People's Hospital
Locations (4):
- China (4):
  - Peking Union Medical College Hospital, Beijin, Beijin
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Guangzhou Twelfth People's Hospital, Guangzhou, Guangdong
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan

IPD SHARING:
Plan to Share IPD: No
Partial clinicopathological data of participants will be presented in the corresponding manuscript.

REFERENCES:
- [Background] Zhang C, Li SL, Nie Q, Dong S, Shao Y, Yang XN, Wu YL, Yang Y, Zhong WZ. Neoadjuvant Crizotinib in Resectable Locally Advanced Non-Small Cell Lung Cancer with ALK Rearrangement. J Thorac Oncol. 2019 Apr;14(4):726-731. doi: 10.1016/j.jtho.2018.10.161. Epub 2018 Nov 5. PMID 30408570
- [Background] Leonetti A, Minari R, Boni L, Gnetti L, Verze M, Ventura L, Musini L, Tognetto M, Tiseo M. Phase II, Open-label, Single-arm, Multicenter Study to Assess the Activity and Safety of Alectinib as Neoadjuvant Treatment in Surgically Resectable Stage III ALK-positive NSCLC: ALNEO Trial. Clin Lung Cancer. 2021 Sep;22(5):473-477. doi: 10.1016/j.cllc.2021.02.014. Epub 2021 Feb 24. PMID 33762169
- [Background] Zhang C, Yan LX, Jiang BY, Wu YL, Zhong WZ. Feasibility and Safety of Neoadjuvant Alectinib in a Patient With ALK-Positive Locally Advanced NSCLC. J Thorac Oncol. 2020 Jun;15(6):e95-e99. doi: 10.1016/j.jtho.2019.12.133. No abstract available. PMID 32471573
- [Background] Chaft JE, Dagogo-Jack I, Santini FC, Eng J, Yeap BY, Izar B, Chin E, Jones DR, Kris MG, Shaw AT, Gainor JF. Clinical outcomes of patients with resected, early-stage ALK-positive lung cancer. Lung Cancer. 2018 Aug;122:67-71. doi: 10.1016/j.lungcan.2018.05.020. Epub 2018 May 22. PMID 30032847
- [Background] Shaw AT, Bauer TM, de Marinis F, Felip E, Goto Y, Liu G, Mazieres J, Kim DW, Mok T, Polli A, Thurm H, Calella AM, Peltz G, Solomon BJ; CROWN Trial Investigators. First-Line Lorlatinib or Crizotinib in Advanced ALK-Positive Lung Cancer. N Engl J Med. 2020 Nov 19;383(21):2018-2029. doi: 10.1056/NEJMoa2027187. PMID 33207094